CLINICAL TRIAL: NCT07227844
Title: Pilot Study of a Mixed-Reality Visual Attention Task for Neglect Diagnosis and Rehabilitation
Brief Title: Mixed-Reality Visual Attention Task for Neglect Diagnosis and Rehabilitation
Acronym: Neglex01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Markey Olson (Other)
Responsible Party: Sponsor-Investigator, Markey Olson, Research Manager, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26-500-131-30-06
Record Dates: First submitted 2025-11-07; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Neglect, Sensory; Neglect, Hemispatial; Neglect, Hemisensory
Keywords: neglect
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: VR Neglect Training

INTERVENTIONS:
Device: VR Neglect Training — VR Neglect Training

SUMMARY:
Neglect, a common and disabling neurological deficit post-CNS injury, profoundly hinders recovery and escalates healthcare costs. Current diagnostic tools are often insensitive or impractical, and while therapies exist, a significant research gap remains. Traditional methods, including standardized scales and paper-pencil tests, lack precision; even advanced video oculography is limited by cost and accessibility. Rehabilitative approaches like visual scanning and prism adaptation offer some benefit, but more effective solutions are needed. This project utilizes a non-invasive neuromodulatory training approach via a mixed-reality visual attention task delivered through a virtual reality headset. This system aims to improve both neglect diagnosis and personalized therapeutic intervention. The study will assess the headset's safety and practicality, its capacity to detect and lateralize neglect, and its long-term effect on improving attention to the neglected field. By measuring reaction times to visual stimuli within the VR environment, the research seeks to develop a more accessible and impactful tool for both assessing and treating neglect, potentially enabling self-directed therapy and enhancing patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The study will involve patients over the age of 18 who have been diagnosed with a neurological injury that includes: ischemic stroke, hemorrhagic stroke, tumor, or trauma.
* Neurological injury that localizes to only one side of the brain
* At least one hand that retains dexterity enough to use a controller to extinguish the visual stimulus.
* Cognitive ability to understand simple instructions on how to use the device
* Visual fields intact

Exclusion Criteria:

* Bilateral symptomatic injury
* Inability to consent or to comply with study
* Blindness or severe visual deficits other than neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Neglect | 6 months
  Measured as improvement in percentage of lines detected at each location in the VR app

SECONDARY OUTCOMES:
Feasibility/Usage, sessions | 6 months
  Number of sessions completed by each participant
Feasibility/Usage, time | 6 months
  Total time spent using the device

CONTACTS AND LOCATIONS:
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided